CLINICAL TRIAL: NCT06591325
Title: Twelve Weeks of Resistance Training is Equally As Effective At Improving Cardiovascular Risk Factors in Older Women with and Without Depression: a Non-randomized Cross-over Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Edilson Serpeloni Cyrino, PhD, Universidade Estadual de Londrina
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GEPEMENE 2024
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depressive Symptoms; Aging; Resistance Training; Cardiovascular Risk Factor
Keywords: strength training; depressive symptoms; anxiety symptoms; cardiovascular risk factor
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise group = participants performed 12 weeks of strength training (Experimental)
  Interventions: Other: exercise; Other: Control
- control group = participants maintained their usual activities normally (No Intervention)

INTERVENTIONS:
Other: exercise — The RT program was performed in the morning and in groups, three days per week (Mondays, Wednesdays, and Fridays), in the University fitness facility over 12 weeks. Participants were personally supervised by Physical Education professionals (1-2 supervisors per exercise session) with substantial RT experience to ensure consistent and safe exercise performance. Throughout the intervention period, the RT program was carried out on machines and free weights (Ipiranga Fitness, Presidente Prudente, SP, Brazil). The training program was carried out in groups. Participants performed four exercises for the trunk and upper limbs (chest press, seated row, triceps pushdown, preacher curl) and four exercises for the lower limbs (horizontal leg press, leg extension, lying leg curl, seated calf raise) in three sets of 10-15 repetitions based on previous guidelines (9,22).
  Arms: exercise group = participants performed 12 weeks of strength training
Other: Control — maintaining the daily routine
  Arms: exercise group = participants performed 12 weeks of strength training

SUMMARY:
Background: the purporse was to evaluate and compare the effects of 12 weeks of resistance training (RT) on cardiovascular disease (CVD) risk factors in older women with and without depressive disorders Methods: We included 79 older women, 52 without depressive disorders and 27 with a diagnosis of depressive disorders. The 79 participants passed through 12 weeks of control condition and were instructed to maintain their habitual routine. After the control period, the participants were reevaluated and attended 12 weeks of RT. The Beck Anxiety Inventory (BAI) and Patient Health Questionnaire-9 (PHQ-9) were used to measure anxiety and depressive symptoms, respectively. The serum levels of high-sensitivity C-reactive protein, glucose, total cholesterol (TC), high-density lipoprotein cholesterol (HDL-c), low-density cholesterol (LDL-c), and triglycerides (TG) were used as cardiovascular risk factors. The Linear Mixed Model (LMM) was used to compare between groups.

DETAILED DESCRIPTION:
1. Introduction It is estimated that 3.8% of the worldwide population (5,7% of adults older than 60 years) experienced a depressive disorder diagnosis in 2023 (1). Further, depression is about 50% more common among women than men. Depressive disorders represent a huge burden for society, especially considering their association with the development of cardiometabolic risk factors and cardiovascular diseases (CVD) (2,3). For instance, several studies found that people with depressive disorders have a higher risk of developing diabetes, metabolic syndrome, CVDs, higher CVD mortality, and all-cause mortality (4,5). Therefore, depressive disorders increase healthcare costs (6), health service utilization (7), and reduce productivity (8). Thus, CVD is the main potentially avoidable contributor to early deaths in patients with depression (4).

   Among the multiple strategies, physical activity is a modifiable behavior that may act as adjuvant therapy for depressive disorders and an essential protective factor for cardiometabolic risk factors and CVD, mainly in older adults (9-11). In this regard, resistance training (RT) has been widely recommended for this population due to its positive impact on overall health and, mainly, to counteract the age-related decline in skeletal muscle mass and muscular strength (9). Particularly, effects of RT has positive effects on cardiometabolic parameters (12,13), body fat (14), cardiorespiratory fitness (15), central nervous system (16), and CVD (14).

   Beyond the benefits for physical health, some systematic reviews and meta-analyses also showed that RT can be effective in reducing depressive and anxiety symptoms in older adults (10,17,18). Additionally, it seems that different clinical conditions (i.e., with vs. without depressive disorders) could present different responses to an RT program, as the participants with depressive disorders presented a higher reduction in depressive symptoms compared with their counterparts (10). This finding indicates that RT may be an effective and feasible intervention for older adults with depressive disorders. Therefore, besides cardiovascular benefits, RT could also be an essential way to protect physical health among people with depressive disorders. However, to our knowledge, there is a lack of studies investigating the effect of RT on CVD risk factors among people with depressive disorders. In addition, depression may impact traditional CVD risk factors such as diet, exercise, as well as adherence to medical treatment aimed at primary and secondary prevention of cardiovascular disease (19). Furthermore, a previous study has shown the association between antidepressant medication and prevalence and poorer control of CVD risk factors in a population-based older adults sample (20). Further, whilst it is generally known that RT can improve CVD in the general population (21), it is unclear if RT is equally effective in those with depression.

   Given the aforementioned, the investigators aimed to evaluate the effects of 12 weeks of RT on CVD risk factors and anxiety and depressive symptoms among older women with and without depressive disorders. Second, the investigators compared the effects of RT on CVD risk factors and anxiety and depressive symptoms among older women with and without depressive disorders. The investigators hypothesized that older women with depressive disorders could have a greater magnitude of improvement in CVD risk factors, anxiety, and depressive symptoms than older women without depressive disorders due to their worse clinical condition.
2. Methods 2.1. Experimental Design

This current investigation is a secondary analysis of the Active Aging Longitudinal Study, designed to analyze the effects of supervised, structured, and progressive RT programs on neuromuscular, morphological, physiological, metabolic, behavioral, and cognitive outcomes in older women. It was selected data collected between November 2021 and July 2022 for the present investigation. This trial was a non-randomized cross-over trial conducted over 33 weeks and divided into two phases:

1. Phase 1 (12 weeks of control condition). One hundred five older women were interviewed, and 79 were selected, from which 27 reported previous medical diagnoses of depressive disorders, while the other 52 participants were free of depressive disorders. Therefore, the 79 participants passed through 12 weeks of control condition and were instructed to maintain their habitual routine (Control Group without Depressive Disorders, n = 52; Control Group with Depressive Disorders, n = 27).
2. Phase 2 (12 weeks of RT). After the control period, the participants were reevaluated and started 12 weeks of RT. Five participants dropped out of the experiment during the follow-up period (three participants without depressive disorders and two participants with depressive disorders). The dropout rate was 5.7% in participants without depressive disorders and 7.4% in participants with depressive disorders. Thus, the final sample of this period consisted of 74 older women (Training Group with Depressive Disorders, n = 25; Training Group without Depressive Disorders, n = 49). Figure 1 shows the flowchart and timeline of this study.

Mental health-related questionnaires (BAI and PHQ-9), biochemical analysis (lipid profile, glucose, and C-reactive protein), and muscular strength tests (1-RM) were performed before the control period, between the control and intervention periods (i.e., post-control and pre-intervention), and after the intervention (weeks 1-3 and 16-18, 31-33) (Figure 1).

2.2. Participants The volunteers were recruited through local TV, radio, newspaper announcements, and social media (WhatsApp, Facebook, and Instagram). Participants completed detailed health history questionnaires and were subsequently admitted to the study if they met the following inclusion criteria: (a) females aged > 60 years; (b) physically independent; (c) had no cardiac, orthopedic, or musculoskeletal dysfunction that could impede physical exercise; (d) not having uncontrolled diabetes mellitus or hypertension; (e) not be involved in the practice of regular physical activity performed more than once a week over the three months before the start of the study; (f) present the medical clearance from a cardiologist (resting 12-lead electrocardiogram test, personal interview, and treadmill stress test when deemed necessary) to attend RT without restriction. To identify participants with depressive disorders, we made an anamnesis where it was asked if the participant had a previous diagnosis of depressive disorders issued by a medical doctor or psychologist and is undergoing treatment for depressive disorders. Participants signed a written informed consent after receiving a detailed description of the investigation procedures. This study was conducted according to the Declaration of Helsinki and approved by the Local Ethics Committee.

2.3. Resistance training program The RT program was performed in the morning and in groups, three days per week (Mondays, Wednesdays, and Fridays), in the University fitness facility over 12 weeks. Participants were personally supervised by Physical Education professionals (1-2 supervisors per exercise session) with substantial RT experience to ensure consistent and safe exercise performance. Throughout the intervention period, the RT program was carried out on machines and free weights (Ipiranga Fitness, Presidente Prudente, SP, Brazil).

The training program was carried out in groups. Participants performed four exercises for the trunk and upper limbs (chest press, seated row, triceps pushdown, preacher curl) and four exercises for the lower limbs (horizontal leg press, leg extension, lying leg curl, seated calf raise) in three sets of 10-15 repetitions based on previous guidelines (9,22). The participants were instructed to inhale during the eccentric phase and exhale during the concentric phase while maintaining a constant movement velocity at a ratio of approximately 1:2 s (concentric and eccentric muscle actions, respectively). Rest intervals were 1-2 and 2-3 min between sets and exercises. The training load was individually adjusted for each exercise weekly, according to the number of repetitions performed during the last training session, to ensure that the subjects kept performing at the ideal intensity for the repetition zone. When participants completed the upper limit of repetitions in all sets for two consecutive sessions, the weight was increased by 2%-5% for the upper limb exercises and 5%-10% for the exercises of the lower limbs 17.

2.4. Primary Outcomes

2.4.1. Cardiovascular risk factors Blood sample (venous) was collected in a tube containing a dipotassium ethylenediaminetetraacetic acid (12 ml, vacuum-sealed system; Vacutainer, England) between 7:00 and 9:00 a.m. by a trained laboratory technician after an overnight fast of at least 12 h. Participants rested in a seated position for at least five minutes before withdrawing 5 ml of blood from a prominent superficial vein in the antecubital space. All samples were centrifuged at 3,000 rpm for 15 min, and plasma or serum aliquots were stored at -80° C until assayed. As determined in human plasma, inter- and intra-assay coefficients of variation were < 10%. Measurements of serum levels of high-sensitivity C-reactive protein, glucose, total cholesterol (TC), high-density lipoprotein cholesterol (HDL-c), and triglycerides (TG) were determined by standard methods in a specialized laboratory at University Hospital. The low-density lipoprotein cholesterol (LDL-c) was calculated using the following equation (23): LDL-c = TC - (HDL-c + TG/5). The analyses were performed using a Dimension RxL Max biochemical auto-analyzer system (Siemens Dade Behring, Erlangen, Germany) according to established methods in the literature consistent with the manufacturer's protocol.

2.5. Secondary Outcomes

2.5.1. Depressive and anxiety symptoms Depressive and anxiety symptoms were assessed using two self-administered questionnaires: the Patient Health Questionnaire (PHQ-9)(24) and the Beck Anxiety Inventory (BAI) (25), respectively. The PHQ-9 consists of nine questions regarding the presence and frequency of depressive symptoms during the previous two weeks. The nine symptoms consist of depressed mood, anhedonia (loss of interest or pleasure in doing things), sleep problems, tiredness or lack of energy, change in appetite or weight, feelings of guilt or worthlessness, problems concentrating, feeling of sluggishness or restlessness, and suicidal thoughts. The frequency of each symptom is assessed on a Likert scale from 0 to 3, corresponding to the answers "never", "several days", "more than half the days" and "almost every day", respectively. The BAI comprises 21 items (statements) about different anxiety symptoms with a 4-point Likert scale, with the final score ranging from 0 to 63. Each item has four possible answers with scores from 0 to 3: 0 = Not at all; 1 = Mild, but it didn't bother me much; 2 = Moderate, it wasn't pleasant at times; 3 = Severe, it bothered me a lot.

2.5.2. Muscular strength Maximal dynamic strength was evaluated using one-repetition maximum (1RM) tests on the leg extension exercise (Ipiranga Fitness, Presidente Prudente, SP, Brazil), respectively, following standard procedures (26). Three 1RM testing sessions were performed over the morning, separated by 48-hour intervals. In each session, participants completed a warm-up of 10-15 repetitions with approximately 50% of the estimated load to the first attempt, followed by three maximal attempts. For the first day of testing, the first selected load was based on the researchers' experience and perception of the difficulty (effort) with which participants performed the warm-up. If the first attempt was completed, the load was added for subsequent attempts (3-10% of the previous effort). If an attempt was unsuccessful, the load was removed in the same proportion. The rest period was three to five minutes between attempts. The load for the first attempt in the second and third sessions was the maximal obtained in the previous session. During each effort, participants were encouraged to perform two repetitions with the selected load. The 1RM was recorded as the heaviest load lifted in one voluntary muscle action among the three sessions. Two experienced researchers supervised all testing sessions to standardize technique reliability and ensure the safety of participants. The standard error of measurement (SEM) and intraclass correlation coefficient (ICC) were satisfactory (SEM = 2.0 kg; ICC = 0.97).

2.6. Characteristics of the sample and potential confounders Age was assessed and presented continuously. Body mass was measured to the nearest 0.1 kg using a calibrated electronic scale Balmak (Laboratory Equipment Labstore, Curitiba, PR, Brazil). Height was measured with a stadiometer attached to the scale to the nearest 0.1 cm. All participants wore light workout clothing and no shoes during the measurements. Body mass index (BMI) was calculated as body mass in kilograms divided by the square of height in meters (27). The Brazilian version of the MoCA was used to analyze the global cognitive function. The MoCA is a screening tool composed of 12 individually punctuated tasks grouped into eight different cognitive domains. The total score ranges from 0 to 30 (higher values reflect better cognition). MoCA psychometric proprieties indicate a high sensitivity (81%) and specificity (77%) for detecting mild cognitive impairment (MCI) states in Brazilian older individuals (28).

2.7. Statistical analysis It was used values of mean and standard deviation as well as relative frequency to describe the characteristics of the sample. Potential differences between the groups during the baseline were assessed using chi-square (categorical variables), Kruskal-Wallis, and one-way ANOVA (continuous variables). The values of pre- and post-control and RT groups were described using mean and standard deviation. It was used linear mixed models to estimate the effect of the RT intervention among the participants with and without depressive disorders by adding an interaction term between time (i.e., pre and post) and group (control and RT), including the participant as a random level. The investigators also used linear mixed models (LMM) to compare the RT intervention effectiveness among participants with and without depressive disorders, adding an interaction term between time and group. The effect size (ES) was calculated as the post-training mean minus the pretraining mean, divided by the pooled pretraining SD (34). An ES of 0.00-0.19 was considered trivial; 0.20-0.49, small; 0.50-0.79, moderate; and ≥0.80, large 24. The statistical analyses were conducted using the software JAMOVI, version 2.4.11 (JAMOVI project, Sydney, AU) and significance was accepted at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* females aged > 60 years;
* physically independent;
* had no cardiac, orthopedic, or musculoskeletal dysfunction that could impede physical exercise;
* not having uncontrolled diabetes mellitus or hypertension;
* not be involved in the practice of regular physical activity performed more than once a week over the three months before the start of the study;
* present the medical clearance from a cardiologist (resting 12-lead electrocardiogram test, personal interview, and treadmill stress test when deemed necessary) to attend RT without restriction.

Exclusion Criteria:

* not reaching 85% of training sessions

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 79 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk factors | From begining to the end 12 weeks
  Blood sample (venous) was collected in a tube containing a dipotassium ethylenediaminetetraacetic acid (12 ml, vacuum-sealed system; Vacutainer, England) between 7:00 and 9:00 a.m. by a trained laboratory technician after an overnight fast of at least 12 h. Participants rested in a seated position for at least five minutes before withdrawing 5 ml of blood from a prominent superficial vein in the antecubital space. All samples were centrifuged at 3,000 rpm for 15 min, and plasma or serum aliquots were stored at -80° C until assayed. As determined in human plasma, inter- and intra-assay coefficients of variation were < 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Undecided